CLINICAL TRIAL: NCT02017769
Title: Magnetic Resonance Imaging and Ultrasound Imaging of Peripheral Nerves in Patients Treated With Immunoglobulin in Chronic Inflammatory Demyelinating Polyradiculoneuropathy.
Brief Title: MRI in Diagnosing and Monitoring CIDP
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-100
Record Dates: First submitted 2013-12-06; First posted 2013-12-23 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Subcutaneous immunoglobulin; Magnetic resonance imaging
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CIDP - treated: Patients diagnosed with CIDP and fulfilling the criteria by EFNS and PNS and in maintenance treatment with subcutaneous immunoglobulin
- Healthy controls: Healthy, gender and age matched controls
- CIDP - untreated: Patients newly diagnosed with CIDP and untreated are treated with immunoglobulin and re-examined after 4 months of treatment

SUMMARY:
We want to study whether MRI can be useful in diagnosing and monitoring patients with CIDP in maintenance treatment with immunoglobulin

DETAILED DESCRIPTION:
Chronic inflammatory neuropathies such as chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) can be successfully treated with immunoglobulin either intravenously (IVIG) or subcutaneously (SCIG).

CIDP is diagnosed by electrophysiology which is time-consuming and unpleasant for the patient.

New techniques suggest that Magnetic Resonance Imaging (MRI) and ultrasound imaging can be used to detect injuries in the peripheral nerves

We want to study if MRI and ultrasound is able to detect damages in peripheral nerves, nerve roots and plexus in patients with CIDP.

Moreover, we want to compare these findings to healthy matched controls and to see if treatment with immunoglobulin changes findings in MRI

ELIGIBILITY:
Inclusion Criteria:

CIDP patients

* Age > 18 and < 80 years
* Diagnosed with definite and probable CIDP and fulfilling the European Federation of Neurological Sciences/Peripheral Nerve Society (EFNS/PNS) criteria

Healthy controls

* Age > 18 and < 80 years
* No neurological disorders

Exclusion Criteria:

* Age < 18 or > 80 years
* Contraindications to MRI
* Pregnancy
* Other cause of neuropathy (incl. pressure neuropathy)
* Diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with subcutaneous immunoglobulin for CIDP are invited to participate. They will be recruited from the outpatient clinic at Department of Neurology in Aarhus, Odense and at Rigshospitalet (Copenhagen)
  Healthy controls will be recruited by public announcement
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
DTI changes in nerves and muscles | At enrolment
  Diffusion Tension Imaging (DTI) in peripheral nerves and muscles in the lower extremities in CIDP patients treated with SCIG will be compared to healthy controls

SECONDARY OUTCOMES:
Changes in MRI findings between treated and untreated CIDP patients | All patients are examined at enrolment. Untreated patients are re-examined after 4 months of treatment
  Comparing changes in MTR and DTI between CIDP patients treated with subcutaneous immunoglobulin to those untreated.
  The untreated patients will be examined again after 4 months of treatment with immunoglobulin
Comparing clinical findings to MRI | At enrolment
  Clinical evaluation by:
  Isokinetic dynamometry Clinical MRC score
  These findings wil be compared to findings on MRI to assess an eventual correlation

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Prof, DMSc, Principal Investigator
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Denmark